CLINICAL TRIAL: NCT05850338
Title: Determination of the Effects of Autogenic Relaxation Exercise and Cold Pillow Application on Vasomotor Symptom Control and Quality of Life in Postmenopausal Women
Acronym: Vasomotor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aylin Güneş (Other)
Responsible Party: Sponsor-Investigator, Aylin Güneş, Asistant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AGunes
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Vasomotor Symptoms; Quality of Life
Keywords: vasomotor symptoms, quality of life
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The data of the study were entered by a person other than the researcher. Statistical analysis was performed by a person other than the researcher. Blinding was done during the evaluation of the data. Intervention and control groups were coded as 1 and 2. The analysis of the data coded in terms of groups was made by the statistician. After the statistical analysis, the coding for the intervention and control groups was explained. Statistical bias was controlled by this blanking technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): the autogenic relaxation exercise would be performed to intervention group. In the first interview, the introductory characteristics form was filled and the Menopause Specific Quality of Life Scale was completed. In addition, women were given training in line with the training booklet about the menopause period, autogenic relaxation exercise and cold pillow. After the training, autogenic relaxation exercise was taught accompanied by the autogenic relaxation exercise CD. The woman was informed about performing autogenic relaxation exercises 3 times a day and using a cold pillow when she experienced vasomotor symptoms. The autogenic relaxation exercise and cold pad application follow-up chart, which was prepared for the purpose of recording the applications, was given. The women were evaluated by being invited to the hospital at 4 and 8 weeks, and they filled out the Menopause Specific Quality of Life Scale during the follow-ups. The intervention was implemented for 8 weeks.
  Interventions: Device: cold pad pillow; Behavioral: autogenic training
- Control (No Intervention): After the women to be included in the control group were determined, individual interviews were conducted with the women in a separate room for orogenic relaxation. In the first interview, the introductory characteristics form was filled and the Menopause Specific Quality of Life Scale was completed. The women were evaluated by being invited to the hospital at 4 and 8 weeks, and they filled out the Menopause Specific Quality of Life Scale during the follow-ups. The women were followed for 8 weeks. No other intervention was applied to the women other than the standard care they received at the hospital. The women were called every week and their vasomotor symptoms were questioned.

INTERVENTIONS:
Device: cold pad pillow — cold pad pillow application when women have vasomotor symptoms for 8 weeks
  Arms: Experimental
Behavioral: autogenic training — Autogenic relaxation for three times a day for eight weeks
  Arms: Experimental

SUMMARY:
The aim of this study was to determine the effect of autogenic relaxation exercise and cold pillows on vasomotor symptom control and quality of life. This randomized controlled study was carried out at Kirikkale University Faculty of Medicine Hospital, Department of Obstetrics and Gynecology, Gynecology Department between 22.06.2018 and 02.01.2019. The sample of the study consisted of 88 people, 44 in the intervention group and 44 in the control group. Since there were case losses in the research, the research was completed with a total of 69 people, 34 in the intervention group and 35 in the control group. The women in the intervention group performed autogenic relaxation exercises and cold pillow application for 8 weeks, and the women in the control group received outpatient care in the hospital. Research data were collected using Descriptive Characteristics Form, Menopause-Specific Quality of Life Scale, Vasomotor Symptom and Practice Follow-up Diary. Data collection tools were applied to the women during the first interview, and at the 4th and 8th weeks after the women were included in the study. In the analysis of descriptive data; number, percentage, mean and standard deviation were used. Independent groups t test was used to determine the difference between groups. The relationship between two independent categorical variables was analyzed using the chi-square test. Variables between dependent groups were compared in repeated measurements with anova test and mixed anova test

DETAILED DESCRIPTION:
Aims:The aim of this study was to determine the effect of autogenic relaxation exercise and cold pillows on vasomotor symptom control and quality of life.

Hypothesis:H0-1: In the postmenopausal period, there was no difference in the frequency of vasomotor symptoms between the group that received autogenic relaxation exercise and cold pillows and the control group.

H1-1: In the postmenopausal period, there is a time difference in vasomotor symptom frequency between the autogenic relaxation exercise and cold pillow group and the control group.

H0-2: In the postmenopausal period, there was no difference in vasomotor symptom duration between the group that was applied autogenic relaxation exercise and cold pillow and the control group.

H1-2: In the postmenopausal period, there is a time difference in vasomotor symptom duration between the autogenic relaxation exercise and cold pillow group and the control group.

H0-3: In the postmenopausal period, there was no difference in vasomotor symptom severity between the groups that received autogenic relaxation exercise and cold pillows and the control group.

H1-3: In the postmenopausal period, there is a time difference in vasomotor symptom severity between the autogenic relaxation exercise and cold pillow group and the control group.

H0-4: In the postmenopausal period, there was no difference in quality of life between the group that was applied autogenic relaxation exercise and cold pillow and the control group.

H1-4: In the postmenopausal period, there is a time difference in quality of life between the group that received autogenic relaxation exercise and cold pillows and the control group.

Design: A parelel design randomised controlled study was conducted according to the CONSORT 2010 guidelines.

Methods: This study was conducted in Kirikkale University Faculty of Medicine Hospital, Department of Obstetrics and Gynecology, Kirikkale, Turkey between 22.6.2018-02.01.2019. The sample of the study consisted of women who were in the postmenopausal period, who met the inclusion criteria and who volunteered to participate in the study.

Inclusion criteria in the study: Being in the first 5-year period of postmenopause, experiencing vasomotor symptoms at least twice a day, being at least literate, living within the borders of the center of Kırıkkale province, not having a disease that mimics vasomotor symptoms, not taking hormone therapy other than estrogen in the last 12 months, not using antidepressants and anxiolytics in the last 3 months, not using herbal alternative treatment within the last 4 weeks, women who do not use other alternative and complementary treatment methods, who have a body mass index below 35 and who do not use hormone replacement therapy.

Sample: A power analysis was utilised to determine the sample size using the G*Power 3.1.7 program. It was calculated that 61 people should be sampled at a significance level of 0.05 for a minimum power of 90%. In order for the number of people in both groups to be equal, 31 interventions were planned to be included in the sample group of 62 people in 31 control groups. In similar studies in the literature, loss of sample during follow-up and since it was seen that there was a sample loss during the preliminary application of our research, it was planned to increase the number of samples by 40% and research groups were formed with 44 people in both groups. 142 women were evaluated in terms of suitability for the study, 45 of the women did not meet the inclusion criteria and 88 women could be included in the study because 9 of them did not agree to participate in the study. At different stages of the study, 10 women from the intervention group and 9 women from the control group withdrew from the study. The research was completed with 34 people in the intervention group and 35 people in the control group. After the research was completed, post-hoc power analysis was performed using the G*power package program and the power of the study was determined as 91% for a sample group consisting of 69 people with a significance level of 0.05 for 34 interventions, 35 control groups and an impact width of 0.225. Intention To Treat (ITT) analysis was performed in the study because there were sample losses.

Randomisation: Since the sample group was not clear before the study, it was recommended that a total of 4 papers, 2 of which were written as "intervention group" and "control group", were thrown into an envelope during the randomization process and that women should be assigned to the relevant group by selecting a paper from this envelope according to the order of participation in the study. The drawn paper was not thrown back into the envelope until the group of four was finished. After the papers in the envelope were finished, the process of assigning women to the relevant groups continued with the same method. After the women pulled the paper from the envelope, they were asked to give it to the researcher without opening the paper. After the women were invited to the study, they were taken to a separate outpatient clinic room and all procedures (randomly assigned to groups, training, teaching autogenic relaxation exercise, etc.) were performed in this room. The women were not told which group they belonged to during the study.

Data collection and outcome measures:The research data were collected using the 'Identifying Features Form', 'Menopause Specific Quality of Life Scale' and 'Vasomotor Symptom and Application Follow-up Diary'.

Introductory features form: In line with the literature were created by researchers with expert opinions. The form includes a total of 28 questions about sociodemographic characteristics, general health status, medical obstetric history and menopausal history.

Menopause-specific quality of life scale: It was developed by Hilditch et al. (1996) to determine the quality of life of women related to menopause and its validity and reliability in Turkish were made by Kharbouch and Şahin (2005). In the Menopause Specific Quality of Life Scale, which consists of 29 items and 4 sub-dimensions, each sub-area score is ranked from 0 to 6. A score of "0" indicates that there is no problem with that issue, a score of "1" indicates that the problem is experienced but not at all, and a score of 2-6 indicates the severity and increasing degrees of the existing problem. The total scale score is not calculated in the Menopause Specific Quality of Life Scale. Scoring is done according to scale sub-dimensions.

Vasomotor symptom and application follow-up diary: It was created by the researchers to record vasomotor symptoms and relaxation exercise and cold pillow application applied in the research by taking expert opinions in line with the literature.

Pilot test: In order to evaluate the intelligibility and usability of the data collection forms, the autogenic relaxation exercise and cold pillow application training booklet and the autogenic relaxation exercise CD to be used in the research, a pre-application was made on 3 women from the intervention and control groups who met the inclusion criteria of the study. Women with pre-treatment were not included in the study sample.

Intervention group: After the women to be included in the intervention group were determined, individual interviews were held with the women in the room where the orogenic relaxation exercise would be performed. A quiet and dim room has been prepared for relaxation exercise. In the first interview, the introductory characteristics form was filled and the Menopause Specific Quality of Life Scale was completed. In addition, women were given training in line with the training booklet about the menopause period, autogenic relaxation exercise and cold pillow. After the training, autogenic relaxation exercise was taught accompanied by the autogenic relaxation exercise CD. The woman was informed about performing autogenic relaxation exercises 3 times a day and using a cold pillow when she experienced vasomotor symptoms. The autogenic relaxation exercise and cold pad application follow-up chart, which was prepared for the purpose of recording the applications, was given. The women were evaluated by being invited to the hospital at 4 and 8 weeks, and they filled out the Menopause Specific Quality of Life Scale during the follow-ups. The intervention was implemented for 8 weeks.

Control group:After the women to be included in the control group were determined, individual interviews were conducted with the women in a separate room for orogenic relaxation. In the first interview, the introductory characteristics form was filled and the Menopause Specific Quality of Life Scale was completed. The women were evaluated by being invited to the hospital at 4 and 8 weeks, and they filled out the Menopause Specific Quality of Life Scale during the follow-ups. The women were followed for 8 weeks. No other intervention was applied to the women other than the standard care they received at the hospital. The women were called every week and their vasomotor symptoms were questioned.

Ethical Approval: Institutional and ethical committee permissions were obtained before starting the study (Approval number: 13/01). In addition, written consent was obtained from the scale owner of the scale to be used in the study and the participants who will participate in the study. After the implementation of the study, the women in the control group were given autogenic relaxation exercise and cold pillow application training and training materials.

Statistical Analysis:Blinding was done during the evaluation of the data. Intervention and control groups were coded as 1 and 2. The analysis of the data coded in terms of groups was made by the statistician. After the statistical analysis, the coding for the intervention and control groups was explained. Statistical bias was checked with this blanking technique.

The research data were transferred to the IBM Statistical Package for Social Sciences (SPSS) 26 program and analyzed. In the study, frequency distributions were used in the evaluation of categorical variables, and descriptive statistics (X̄±SD) were used for numerical variables. The scale sub-dimension scores of the Menopause Specific Quality of Life Scale, which was used as a measurement tool in the research, were obtained by taking the sum of the related items. The mixed-pattern anova test was used to test changes or differences in repeated measures of within-group (in-group effect), between-group (time) effect, and co-effect (group*time effect) repeated measures in intervention and control groups. The margin of error for statistical analysis results was accepted as 5%. In the evaluation of the effect size, the partial η2 value was used (small effect size=0.01, medium effect size=0.06 and large effect size=0.14). The negative (-) value in front of the effect sizes indicates that the initiatives have a negative effect; a positive (+) value indicates that interventions have a positive effect (230).

Intention To Treat (ITT) analysis was performed because there were sample losses in the study. The results of the analyzes (ITT) and Per Protocol (PP) were similar.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing vasomotor symptoms at least twice a day Least literate Living within the borders of Kirikkale province Women who consented to participate in the study

Exclusion Criteria:

* Those with hyperthyroidism, pheomacrocytoma, carcinoid syndrome, diabetes mellitus, cancer, tuberculosis, and other chronic infections (Since the symptoms in these diseases can mimic vasomotor symptoms or the disease may cause hot flashes)

  * Receiving hormone therapy other than estrogen in the last 12 months (as it affects ovarian function and increases the symptoms of hot flashes)
  * Receiving antidepressant and anxiolytic treatment regularly in the last 3 months (because these drugs reduce the symptoms of hot flashes)
  * Receiving herbal alternative treatment in the last 4 weeks (since these treatments have a prolonged effect)
  * Using other alternative and complementary medicine methods (as it may cause errors while evaluating the study results)
  * Having a Body Mass Index of 35 and above
  * Using Hormone Replacement Therapy
  * Women who had a condition that prevented them from using cold pillows (sensory disorder, mental state disorder, circulatory disorder, open wound, cold allergy, hypersensitivity to cold)

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postmenopausal women were included in this study.
Enrollment: 88 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
frequency of vasomotor symptoms number | eight weeks
  vasomotor symptoms experienced per day

SECONDARY OUTCOMES:
vasomotor symptom duration | eight weeks
  duration of vasomotor symptom experienced/minute

OTHER OUTCOMES:
vasomotor symptom severity | eight weeks
  score
menopause-specific quality of life | eight weeks
  menopause-specific quality of life scale was used to evaluate

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Gunes, RN, PhD, Study Chair — Kırıkkale University
Locations (1):
- Aylin Gunes, Ankara, Keçi̇ören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The confidentiality of the data used in the study will be protected.